CLINICAL TRIAL: NCT04082312
Title: Risk Factors and Prognosis of Acute Kidney Injury in Peri Operative Cardiac Surgery Adult Patients Supported by VA-ECMO
Brief Title: Acute Kidney Injury in Adult Patients Supported by VA-ECMO
Acronym: AKI-ECMO
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Adrien Bouglé, Head of Surgical Intensive Care Unit, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: AKI-ECMO
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acute Kidney Injury; Cardiogenic Shock
Keywords: Acute Kidney Injury; ECMO; Post Cardiogenic Shock Syndrome
MeSH Terms: conditions — Acute Kidney Injury; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients admitted in the surgical intensive care unit in post-operative of cardiac surgery between January 2013 and December 2016 + Assisted by VA-ECMO + with KDIGO stage 3 AKI
  Interventions: Other: No intervention
- Group 2: Patients admitted in the surgical intensive care unit in post-operative of cardiac surgery between January 2013 and December 2016 + Assisted by VA-ECMO + without KDIGO stage 3 AKI and alive at D10
  Interventions: Other: No intervention
- Group 3: Patients admitted in the surgical intensive care unit in post-operative of cardiac surgery between January 2013 and December 2016 + Assisted by VA-ECMO + died before D10 without KDIGO stage 3 AKI
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Post-cardiotomy cardiogenic shock (PCCS) occurs in 2-6% of patients undergoing cardiac surgery, and 1% of cardiac surgery patients will require mechanical circulatory support using Veno-Arterial ExtraCorporeal Membrane Oxygenation (VA-ECMO). Acute Kidney Injury is a frequent complication in this population and negatively impacts the survival. We aimed to determine whether the timing of ECMO implantation influence the renal prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in post-operative of cardiac surgery
* Assisted by VA-ECMO

Exclusion Criteria:

* Chronic hemodialysis
* Death occurring within the first 48 hours of VA-ECMO implantation
* Multiple VA-ECMO during the same hospitalization.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the Surgical Intensive Care Unit of the Cardiology Institute of La Pitié Salpêtrière University Hospital (Paris, France) between January 2013 and December 2016.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of a stage 3 AKI | Day 10 after ECMO implantation
  Number of Participants with Stage 3 Acute Kidney Injury according to the Kidney Disease: Improving Global Outcomes (KDIGO) group

SECONDARY OUTCOMES:
Mortality at Day 30 | Day 30 after ECMO implantation
  Number of Deceased Participants
Mortality at 6 months | 6 months after ECMO implantation
  Number of Deceased Participants

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Adrien Bouglé, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lepere V, Duceau B, Lebreton G, Bombled C, Dujardin O, Boccara L, Charfeddine A, Amour J, Hajage D, Bougle A. Risk Factors for Developing Severe Acute Kidney Injury in Adult Patients With Refractory Postcardiotomy Cardiogenic Shock Receiving Venoarterial Extracorporeal Membrane Oxygenation. Crit Care Med. 2020 Aug;48(8):e715-e721. doi: 10.1097/CCM.0000000000004433. PMID 32697513